CLINICAL TRIAL: NCT00564746
Title: A Study to Investigate the Excretion Balance of SB-681323 in Healthy Male Volunteers [Type 3C]
Brief Title: To Assess the Excretion Balance and Pharmacokinetics of a Single Oral Dose of [14C]SB-681323 in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SB681323/011
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: SB-681323,; ADME,; radiolabel
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (1):
- 6 subjects in a single cohort (Experimental): Each subject will be administered a single 10 milligrams (50 microcurie) oral dose of [14C]SB-681323.
  Interventions: Drug: A single 10 milligram (50 microcurie) oral dose of [14C]SB-681323

INTERVENTIONS:
Drug: A single 10 milligram (50 microcurie) oral dose of [14C]SB-681323 — [14C] SB-681323 oral solution, is available as a powder which will be made into a solution of 0.1 milligram/milliliter (0.5 microcurie) [14C] SB-681323 in dextrose and water for injection on the day prior to dosing.
  For a 10 milligram/50 microcurie oral dose of [14C]SB-681323, 100 milliliters of 0.1 milligram/milliliter (0.5 microcurie/milliliter [14C] SB-681323 oral solution will be dosed.

SUMMARY:
SB-681323 is a p38 MAP kinase inhibitor and is currently under development by GlaxoSmithKline. This will be an open label study conducted at one site. Six healthy male subjects will be enrolled to ensure at least four fully evaluable subjects. Each subject will receive a single 10mg/ 50 µCurie oral dose of [14C]SB-681323. Urine and faecal samples will be collected until 216 h after dosing but subjects may be discharged after 168 h if 90% of the dose is recovered and/or <1% of the dose is excreted in a 24 h period. Blood and plasma will be collected at various sample times after dosing to measure parent drug and total drug-related material. Samples of urine, faeces and plasma will be transferred into separate study to characterise and quantify metabolites in these matrices. Safety will be assessed by adverse event monitoring, vital signs, ECG and clinical laboratory tests.

DETAILED DESCRIPTION:
This will be an open label study conducted at one site. Six healthy male subjects will be enrolled to ensure at least four fully evaluable subjects. Each subject will receive a single 10mg/ 50 µCurie oral dose of [14C]SB-681323. Urine and faecal samples will be collected until 216 h after dosing but subjects may be discharged after 168 h if 90% of the dose is recovered and/or <1% of the dose is excreted in a 24 h period. Blood and plasma will be collected at various sample times after dosing to measure parent drug and total drug-related material. Samples of urine, faeces and plasma will be transferred into separate study to characterise and quantify metabolites in these matrices. Safety will be assessed by adverse event monitoring, vital signs, ECG and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged between 30 and 60 years inclusive, at the time of screening.
* Body weight = 50 kg (110 lbs).
* A body mass index (BMI) within the range of 18.5 to 29.9 kg/m2 inclusive.
* Signed and dated written informed consent prior to admission to the study.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination, or ECG (12-lead).
* Significant cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal conditions that in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as participant in this trial.
* QTc(b) > 450msecs
* A definite or suspected personal or family history of adverse reactions or hypersensitivity to the trial drug or to drugs with a similar chemical structure.
* History of regular alcohol consumption exceeding an average weekly intake of > 21 units (or an average daily intake of greater than 3 units). One unit is equivalent to a half-pint (284mL) of beer/lager; 25mL measure of spirits or 125mL of wine).
* Subjects with a history or presence of gastro-intestinal or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Subjects who have consumed grapefruit or grapefruit juice within seven days of the first study day.
* Subjects who have had exposure to more than three new chemical entities within 12 months prior to the first dosing period.
* Subjects who have participated in a trial with a different new chemical entity within 90 days prior to the start of this study.
* If participation in the study will result in the volunteer having donated more than 400mL of blood in the previous 56 days.
* Subjects who have received a total body radiation dose of greater than 5.0 mSv (upper limit of WHO category II) or exposure to significant radiation (e.g. serial Xray or CT scans, barium meal etc) in the 12 months prior to this study.
* History of elevated blood pressure or blood pressure persistently >140/90 mmHg at screening.
* An unwillingness to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness of the subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, sub-dermal implants or a tubal ligation if the women could become pregnant from the time of the first dose of the study medication until completion of the follow-up procedures.
* Lack of suitability for participation in this study, for any reason, in the opinion of the investigator.
* Any condition that could interfere with the accurate assessment and recovery of 14C.

Prescribed or over-the-counter medication within 5 days (or 5 half lives, whichever is longer) prior to the first dosing day, unless the investigator confirms that it will not introduce additional risk or interfere with the study procedures or outcome.

* Liver function tests (ALT, AST, ALP, ?GT and bilirubin) > upper limit of normal (ULN) at screening
* Creatinine phosphokinase (CPK) > ULN at screening
* Positive urine drug screen
* Positive HIV, Hepatitis B or C result at screening.
* History of use of tobacco- or nicotine-containing products within 6 months of screening or a positive urine cotinine screen (urine cotinine > 250ng/mL).

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2007-09-20 (Actual); Primary Completion 2007-10-26 (Actual); Study Completion 2007-10-26 (Actual)

PRIMARY OUTCOMES:
Urinary and faecal cumulative excretion as a percentage of the total radioactive dose administered over time. | 168 Hours

SECONDARY OUTCOMES:
AUC(0-8), Cmax, AUC(0-t), tmax and t½ of total radioactivity and SB8681323 in plasma following oral dosing.- Blood:Plasma ratio of total radioactivity.- AEs, ECG, vital signs and clinical laboratory tests (including LFTs). | 216 Hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tranent, West Lothian, United Kingdom

REFERENCES:
- See also: Results for study 681323/011 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/SB681323/011?search=study&search_terms=681323%2F011#rs